CLINICAL TRIAL: NCT07405580
Title: THE EFFECT OF A PREPARATİON PROGRAM FOR CLİNİCAL PRACTİCE BASED ON THE EXCELLENCE MODEL ON STUDENTS' READİNESS, EXCELLENCE, CLİNİCAL COMFORT, AND ANXİETY LEVELS: A RANDOMİZED CONTROLLED TRİAL
Brief Title: THE EFFECT OF A CLINICAL PRACTICE PREPARATION PROGRAM BASED ON THE EXCELLENCE MODEL ON STUDENTS: A RANDOMIZED CONTROLLED TRIAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Öğr. Gör. Hamide COŞKUN ERÇELİK, instructor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PAMUKKALEU-COSKUNERCELİK-001
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: This Study Focuses on the Impact of the Pediatric Nursing Excellence Model on Nursing Education
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine orientation training and a clinical practice readiness program based on the excellence model (Experimental)
  Interventions: Other: Educational intervention
- routine orientation training (No Intervention)

INTERVENTIONS:
Other: Educational intervention — In the study, students in the experimental group will undergo a clinical practice preparation program based on the excellence model, unlike those in the control group.
  Arms: routine orientation training and a clinical practice readiness program based on the excellence model

SUMMARY:
Objective: This study was designed to develop a clinical practice preparation program based on the Pediatric Nursing Excellence Model for undergraduate nursing students and to evaluate the program's effect on students' readiness, clinical comfort and anxiety, and levels of excellence.

Method: This study is a pretest-posttest randomized controlled experimental study. The research is planned to be conducted with nursing students taking the Pediatric Health and Disease Nursing course. The study groups will consist of students who go out for clinical practice within the scope of this course. In the power analysis performed with the G*Power 3.1.9.7 program, the sample size was found to be 25 for the experimental group and 25 for the control group, for a total of 50. Research data will be collected using a questionnaire. The questionnaire consists of four sections containing the following questions: "Student Descriptive Characteristics Information Form," "Nursing Students' Readiness for Clinical Practice Scale," "Pediatric Nursing Students' Clinical Comfort and Anxiety Instrument," and "Pediatric Nursing Excellence (PHM) Model Questionnaire." In the study, students in the experimental group will receive routine orientation training and a clinical practice readiness program based on the excellence model. Students in the control group will only receive routine orientation training. Data analysis will be performed using the SPSS 20.0 software package.

ELIGIBILITY:
Inclusion criteria:

* Being a nursing student,
* Taking the Child Health and Nursing course for the first time,
* Attending the course,
* Not having previously taken pediatric nursing readiness training,
* Agreeing to participate in the study voluntarily.

Exclusion criteria:

* The student's refusal to participate in the study,
* Withdrawal from the study before completing all stages of the research.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2026-06-16 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Students' Readiness Levels for Clinical Practice | [Time Frame: one day in the first week of clinical practice] [Time Frame: one day in the third week of clinical practice] [Time Frame: one day in the last week (seventh) of clinical practice]
  The assessment will be conducted using the 'Clinical Readiness Scale' developed by Avşar et al. (2024). The scale consists of 4 sub-dimensions and a total of 31 items: "Clinical Decision-Making and Application Skills," "Ensuring Safety and Effective Communication," "Basic Knowledge and Holistic Care," and "Understanding the Field of Practice." The scale is scored on a 5-point Likert scale as "strongly disagree (1)", "disagree", "somewhat agree", 'agree', and "strongly agree (5)". The scale is calculated based on the item mean score. The lowest possible score on the scale and its subscales is 1, and the highest possible score is 5. There are no reverse items on the scale. The Cronbach's alpha coefficient for the entire scale was determined to be 0.964. As the score on the scale increases, the level of readiness for clinical practice increases.

SECONDARY OUTCOMES:
Students' Clinical Comfort and Worry | [Time Frame: one day in the first week of clinical practice] [Time Frame: one day in the third week of clinical practice] [Time Frame: one day in the last week (seventh) of clinical practice]
  The 'Pediatric Nursing Students Clinical Comfort and Worry Scale' developed by Arslan et al. (2018) will be used for evaluation. The scale has two subscales: comfort level and worry level. The scale consists of a total of 11 questions, six of which assess students' comfort level during pediatric clinic practice, and five of which assess their worry level. The scale is scored on a 4-point Likert scale as "strongly agree," "agree," "disagree," and "strongly disagree." The third and fifth items in the comfort dimension of the scale are reverse-scored. The Cronbach's alpha coefficient for the comfort dimension of the scale was found to be 0.68, and the Cronbach's alpha coefficient for the worry dimension was found to be 0.89. High scores on the comfort and worry dimensions indicate higher levels of comfort and worry, respectively.
Pediatric Nursing Excellence Level | [Time Frame: one day in the first week of clinical practice] [Time Frame: one day in the third week of clinical practice] [Time Frame: one day in the last week (seventh) of clinical practice]
  Students' levels of excellence in pediatric nursing will be assessed using the "Pediatric Nursing Excellence Model Questionnaire" prepared by the researchers. This questionnaire will be adapted from the original framework of the Pediatric Nursing Excellence (PH) model, which is based on and related to the relevant literature.

CONTACTS AND LOCATIONS:
Overall Officials: SEBAHAT ALTUNDAĞ, Principal Investigator — Pamukkale University

IPD SHARING:
Plan to Share IPD: No